CLINICAL TRIAL: NCT07380295
Title: Improving Workforce Participation and Well-Being in Individuals With Multiple Sclerosis- A Feasability Study
Brief Title: Improving Workforce Participation and Well-Being in Individuals With Multiple Sclerosis - A Feasability Study
Status: Recruiting | Type: Observational
Sponsor: Region Gävleborg (Other)
Collaborators: University of Gavle (Other)
Responsible Party: Sponsor
Other Study IDs: MSCogWork3
Record Dates: First submitted 2025-09-22; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with multiple scleroris of working age: Patients with MS and of working age (18-65) referred to neuropsychological evaluation.

SUMMARY:
Multiple sclerosis (MS) is a chronic neurodegenerative disease and a leading cause of reduced workforce participation due to neurological illness in Western countries. Over the past 30 years, new treatments have reduced symptom burden, allowing patients to stay in the workforce longer. However, fatigue and cognitive impairments remain major barriers to work capacity. This project aims to preliminary examine the impact of cognitive function on work ability, and assess the role of neuropsychologists in multidisciplinary rehabilitation teams. It consists of a feasibility study evaluating the integration of neuropsychological interventions into teambased work-oriented rehabilitation. The specific research questions are:

1. How can neuropsychological interventions be integrated into team-based work-oriented rehabilitation?
2. How do these interventions relate to work ability and well-being in individuals with MS? The investigators plan to collect data on 20 consecutively patients with MS before, 6 months after and 2 years after a neuropsychological testing and intervention. The patients are being followed on measures related to well-being and work ability. Data from the neuropsychological assessment, other rehabilitation interventions as well as data related to treatment and progress of MS are also collected.

Our findings aim to enhance work-oriented rehabilitation and provide a deeper understanding of how to support individuals with MS in maintaining employment and overall well-being

ELIGIBILITY:
Inclusion Criteria:

Multiple sclerosis Age between 18-65 Refered to neuropsychological assessment at the Neurology departement at Gävle Hospital -

Exclusion Criteria:

Other diagnosis hindering work participation more than MS

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of working age with MS in Region Gävleborg who are refered for a neuropsychological assessment and who are not suffering from other diagnosis which impact their work ability to a large extent.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Work participation | From baseline to 2-year follow-up
  Percentage of full-time work. 100 % full-time work and 0% is not working at all.
Hospital anxiety and depression scale | From baseline to 2-year follow-up
  Self-assessment of anxiety and depression. Consists of two scales measuring the probability of having anxiety and depression respectively. Min score 0, max 21 for each scale. Higher scores indicate higher probability of anxiety/depression.
WHO-5 Well-Being Index | From baseline to 2-year follow-up
  Overall rating of well-being. The WHO-5 score range is a raw score of 0-25, which is then multiplied by 4 to get a percentage score of 0-100. Higher score indicates higher well-being.
Brief index of job satisfaction | From baseline to 2-year follow-up
  The Brief Index of Affective Job Satisfaction (BIAJS) has a score range of 1 to 5 for each of its four items, based on a 5-point Likert scale where 1 is "strongly disagree" and 5 is "strongly agree". The total BIAJS score is the sum of these four items, resulting in a possible range from 4 to 20, with higher scores indicating greater affective job satisfaction.

SECONDARY OUTCOMES:
Quantative work demands | From baseline to 2-year follow-up
  Questions from the subscale "Quantitative demands" of the Copenhagen Psychosocial Questionnaire (COPSOQ-III) related to the demands of work. The COPSOQ-III uses Likert-like scales, and its items are coded with values of 0, 25, 50, 75, and 100 to achieve a 0-100 scale. Higher scores indicate more demands.
Can-Work-S | From baseline to 2-year follow-up
  Three questions from a questionnaire developed to measure work-life balance after cancer. Each item ranges from 1 to 5 with higher scores indicating worse work-life balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Gävle hospital, Gävle, Sweden

IPD SHARING:
Plan to Share IPD: No
To comply with the conditions set by the ethical review board, individual participant data (IPD) cannot be shared with other researchers. However, aggregated data are available upon reasonable reques